CLINICAL TRIAL: NCT01198782
Title: Evaluating Safety and Efficacy of FID 112903 Post Discontinuation of Long-term Use of RESTASIS® (Cyclosporine Ophthalmic Emulsion) 0.05%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-42
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FID 112903 (SYSTANE® ULTRA Lubricant Eye Drops) (Experimental): SYSTANE® ULTRA Lubricant Eye Drops dosed 4 times daily
  Interventions: Other: FID 112903 (SYSTANE® ULTRA Lubricant Eye Drops)

INTERVENTIONS:
Other: FID 112903 (SYSTANE® ULTRA Lubricant Eye Drops) — Patients will dose 4 times daily for 4 months.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of FID 112903 given as an immediate treatment replacement in dry eye subjects that discontinue at least 6 months use of RESTASIS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Patients must have a best corrected visual acuity of 0.6 LogMar or better in each eye, and must use Restasis BID for at least 6 months.
* Lastly, patients must have a sodium fluorescein (NaFl) corneal staining sum score of greater than or equal to 3 in the worse eye.

Exclusion Criteria:

* Patients cannot wear contact lenses during the study and cannot have a history of hypersensitivity to any component of FID 112903.
* Patients cannot have ocular or intraocular surgery or serious ocular trauma within the past 6 months, and cannot have punctal plugs of any type.
* Patients cannot use any prescription topical medication for other ocular conditions (such as glaucoma, uveitis, etc).
* Patients cannot use systemic medications that may contribute to dry eye if the dosing regimen has not been stable for at least 30 days prior to Visit 1.
* Patients cannot have ocular conditions that, in the opinion of the investigator, preclude the safe administration of the test article.
* Patients cannot have a history and/or current evidence of the following: epithelial herpes simplex keratitis (dendritic keratitis); vaccinia, active or recent varicella viral disease of the cornea and/or conjunctiva; active ocular rosacea; acute or chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal diseases of the eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The change from baseline in Total Corneal Staining. | 4 months

REFERENCES:
- [Result] http://iovs.arvojournals.org/article.aspx?articleid=2353102